CLINICAL TRIAL: NCT01011959
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Ascending Parallel-group Study of the Safety and Tolerability of REGN88 in Subjects With Rheumatoid Arthritis Receiving Concomitant Methotrexate
Brief Title: A Multiple-dose Study of the Safety and Tolerability of REGN88(SAR153191) in Rheumatoid Arthritis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6R88-RA-0802
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): dose 1 vs. placebo
  Interventions: Biological: REGN88
- 2 (Active Comparator): dose 2 vs. placebo
  Interventions: Biological: REGN88
- 3 (Active Comparator): dose 3 vs. placebo
  Interventions: Biological: REGN88
- 4 (Active Comparator): dose 4 vs. placebo
  Interventions: Biological: REGN88
- 5 (Active Comparator): dose 5 vs. placebo
  Interventions: Biological: REGN88
- 6 (Active Comparator): dose 6 vs. placebo
  Interventions: Biological: REGN88

INTERVENTIONS:
Biological: REGN88 — This study will be conducted in 3 parts, and will include a total of 6 dose cohorts. Part B will not begin until the safety of Part A has been assessed. Part C will begin when enrollment into Part B is complete.

SUMMARY:
This is a randomized study of the safety and tolerability of multiple doses of REGN88 in rheumatoid arthritis patients who are receiving treatment with methotrexate.

DETAILED DESCRIPTION:
This is a multi-centered, randomized, double-blind, placebo-controlled, ascending parallel-group study of the safety and tolerability of REGN88 in patients with rheumatoid arthritis who are receiving concomitant methotrexate.

This study will be conducted in 3 parts, and will include a total of 6 dose cohorts. Part B will not begin until the safety of Part A has been assessed. Part C will not begin until enrollment in Part B is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of Rheumatoid Arthritis
* Patients currently treated with concomitant methotrexate for at least 12 weeks, with a stable dose for at least 6 weeks

Exclusion Criteria:

* Persistent chronic or current active infections
* Patients who have taken anakinra within 2 weeks
* Patients who have taken etanercept, cyclosporine, mycophenolate, tacrolimus, gold, penicillamine, sulfasalazine or hydroxychloroquine within 4 weeks
* Patients who have taken adalimumab within 6 weeks
* Patients who have taken abatacept, azathioprine, cyclophosphamide or infliximab within 12 weeks
* Patients who have taken leflunomide or rituximab within 6 months
* Patients who have had prior treatment with tocilizumab or any other anti-IL-6 medication
* Significant arthritis or other medical condition that could interfere with study evaluations
* Participation in any clinical research study evaluating another investigational drug within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in patients treated with REGN88 and placebo | 10 weeks

SECONDARY OUTCOMES:
To evaluate exploratory efficacy endpoints | over 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allen Radin, MD, Study Director — Regeneron Pharmaceuticals
Locations (24):
- United States (24):
  - Santa Maria, California
  - Boca Raton, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Delray Beach, Florida
  - Palm Harbor, Florida
  - Idaho Falls, Idaho
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Flowood, Mississippi
  - Kalamzaoo, Missouri
  - St Louis, Missouri
  - Reno, Nevada
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Greenville, South Carolina
  - Orangeburg, South Carolina
  - Hixson, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas